CLINICAL TRIAL: NCT05685615
Title: A Multicenter, Open-label, Randomized, Active-controlled, Phase 2 Study to Evaluate the Pharmacokinetics, Efficacy, and Safety of Intravenous BV100 Combined with Polymyxin B Versus Best Available Therapy in Adult Patients with Ventilator-associated Bacterial Pneumonia Suspected or Confirmed to Be Due to Carbapenem-resistant Acinetobacter Baumannii
Brief Title: PK of BV100 in Patients VABP Suspected or Confirmed to Be Due to CRAB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioVersys AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BV100-006
Record Dates: First submitted 2023-01-04; First posted 2023-01-17 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2023-11

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Polymyxin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- BV100 (200 mg) plus Polymyxin B (Experimental): BV100 (200 mg q12h) infused over 2 hours plus Polymyxin B (12 500-15 000 IU/kg) infused over 1h
  Interventions: Drug: BV100 plus Polymyxin B
- BV100 (300 mg) plus Polymyxin B (Experimental): BV100 (300 mg q12h) infused over 2 hours plus Polymyxin B (12 500-15 000 IU/kg) infused over 1h
  Interventions: Drug: BV100 plus Polymyxin B
- Best Available Therapy (Active Comparator): Best Available Antibiotic Therapy to Treat CRAB
  Interventions: Drug: BAT
- Part B: BV100 plus BAT (Experimental): BV100 (300 mg q12h) infused over 2 hours plus Best Avaialble Therapy to Treat Colistin resistant CRAB
  Interventions: Drug: BAT

INTERVENTIONS:
Drug: BV100 plus Polymyxin B — Rifabutin for Infusion plus Polymyxin B for Injection
  Arms: BV100 (200 mg) plus Polymyxin B; BV100 (300 mg) plus Polymyxin B
Drug: BAT — The best avaialble antibiotic therapy to treat CRAB
  Other Names: Best Avaialble Therapy
  Arms: Best Available Therapy; Part B: BV100 plus BAT

SUMMARY:
A multicenter Phase 2 study to evaluate the pharmacokinetics, efficacy, and safety of intravenous BV100 combined with Polymyxin B in adult patients with VABP suspected or confirmed to be due to CRAB

DETAILED DESCRIPTION:
A multicenter, open label, randomized, active controlled, Phase 2 study to evaluate the pharmacokinetics, efficacy, and safety of intravenous BV100 combined with Polymyxin B versus best available therapy in adult patients with ventilator associated bacterial pneumonia suspected or confirmed to be due to carbapenem-resistant Acinetobacter baumannii

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all the following diagnostic and clinical criteria are eligible for the study:

1. Provide written informed consent prior to any study related procedures not part of normal medical care. Surrogate consent/use of a legally authorized representative may be provided, if permitted by local country and institution specific guidelines. If a patient regains consciousness while in the study and, per the Investigator's judgment, the patient is able to read, assess, understand, and make his/her own decision to participate in the trial, the patient can agree to continue participation and the patient should be re consented, if required by local country and institution specific guidelines.
2. Male or female patients ≥ and < 80 years of age at the time of Informed Consent Form (ICF) signing with a body mass index (BMI) of < 40 kg/m2 at the time of ICF signing.
3. Hospitalized for ≥ 48 hours, intubated (via endo or nasotracheal tube, including tracheostomy patients) and receiving mechanical ventilation for ≥ 48 hours at the time of randomization, and with acute changes made in the ventilator support system to enhance oxygenation, as determined by arterial blood gas, or worsening PaO2/FiO2 ratio.
4. All patients must have a chest radiograph or a lung CT scan within 48 hours prior to randomization showing the presence of new or progressive infiltrate(s) suggestive of bacterial pneumonia (based on Investigator's evaluation).
5. Clinical findings to support diagnosis of VABP. At least 1 of the following must be documented to be present within 24 hours prior to randomization:

   * Documented fever (oral ≥ 38.0 °C [100.4 °F] or a tympanic, temporal, rectal, or core temperature ≥ 38.3 °C [101.0 °F], axillary or forehead scanner ≥ 37.5 °C [99.5 °F]) OR
   * Hypothermia (rectal/core body temperature ≤ 35.0 °C [95.2 °F]), OR
   * Leukocytosis with total peripheral white blood cell count (WBC) ≥ 10 000 cells/mm3, OR
   * Leukopenia with total peripheral WBC count ≤ 4500 cells/mm3.
6. Acute Physiology and Chronic Health Evaluation (APACHE II) score between 8 and 30, inclusive, within 24 hours prior to randomization. Any data collected before ICF signature as part of a routine standard for patient care (e.g., laboratory values, Glasgow Coma Score, Acute Physiology Score [APS]) can be used for Screening Visit assessment, if applicable, without repeating the assessments.
7. High probability of pneumonia due to A. baumannii, defined as follows:

   * RDT, performed within 36 hours prior to randomization, using an acceptable respiratory sample (PBS, BAL, mini BAL, or ETA) positive for A. baumannii, OR
   * A surveillance culture from a respiratory sample positive for A. baumannii within 72 hours prior to randomization.

Part B specific:

1. Patients who have been treated previously with an empiric antibiotic regimen and have failed treatment, both clinically and microbiologically, if they have an identified CRAB which has been shown to be non-susceptible in vitro to each of the antibiotic(s) of the empiric antibiotic regimen or has been identified from a culture performed after at least 48 hours of empiric antibiotic regimen, AND/OR
2. Has an infection caused by A. baumannii organisms known to be resistant to colistin (defined as MIC ≥ 4 mg/L by a non-agar-based method) based on evidence from culture or susceptibility testing after at least 48 hours of antibiotic treatment.

Exclusion Criteria:

* Patients who meet any of the following criteria are not eligible to participate in this study:

  1. Known or suspected community acquired bacterial pneumonia or viral, fungal, or parasitic pneumonia.
  2. Sustained shock with persisting hypotension requiring vasopressors to maintain mean arterial pressure ≥ 60 mmHg
  3. Known or suspected allergy to polymyxin, rifabutin, BAT, or their excipients.
  4. Any of the following health conditions:

     * Confirmed legionella infection (Legionella pneumophila pneumonia), Aspergillus spp. pneumonia (testing is not required)
     * Candida spp. infection requiring systemic treatment
     * Cystic fibrosis
     * Known or suspected Pneumocystitis jiroveci pneumonia
     * Known or suspected active tuberculosis
     * Lung abscess
     * Solid organ transplant within 6 months prior to randomization
     * Pleural empyema
     * Evidence of deep seated infection outside the respiratory tract, e.g., endocarditis, osteomyelitis.
     * Known or suspected neuropathy or neuromuscular disease
     * Known HIV infection
  5. Bronchial obstruction or a history of post obstructive pneumonia (this does not exclude patients with pneumonia who have an underlying chronic obstructive pulmonary disease).
  6. Acute graft versus host disease Grade ≥ 3.
  7. Expected survival < 72 hours or a Do Not Resuscitate Order.
  8. Burns > 40% of total body surface area.
  9. Current or anticipated neutropenia with absolute neutrophil count < 1000 cells/mm3.
  10. Severe renal disease defined as an estimated creatinine clearance as per Cockcroft Gault (CLCR CG) < 30 mL/minute or estimated glomerular infiltration rate (eGFR) as per Modified Diet in Renal Disease (MDRD) equation < 30 mL/min/1.73 m2, or requirement for peritoneal dialysis, hemodialysis, hemofiltration, or a urine output < 20 mL/hour over a 24 hour period.
  11. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or bilirubin (conjugated/unconjugated) ≥ 3 × upper limit of normal (ULN) values used by the laboratory performing the test or Child Pugh Class B and C in patients with chronic liver function impairment. Evidence of significant hepatic disease or dysfunction, including known acute viral hepatitis, hepatic cirrhosis, hepatic failure, chronic ascites, or hepatic encephalopathy.
  12. Received systemic or inhaled antibiotic therapy potentially effective against A. baumannii within 72 hours prior to randomization for ≥ 36 hours
  13. Investigator's opinion of clinically significant electrocardiogram (ECG) finding such as new ischemic changes, infarct, or ventricular arrhythmia with immediate potential for a fatal outcome, bradycardia not corrected by pacemaker or medication, or, prior to the current infection, a history of New York Heart Association (NYHA) Class IV cardiac failure defined as severe limitations - experiences symptoms even while at rest, mostly bedbound patients, within 1 year.
  14. Abnormal QT interval corrected by Fridericia (QTcF): > 450 ms confirmed with repeat ECG.
  15. Stroke (ischemic or intracerebral hemorrhage) within 5 days prior to randomization.
  16. Women who are pregnant or nursing, or who are of childbearing potential and unwilling to use an acceptable method of birth control (e.g., intra-uterine device [IUD], male partner sterilization, or complete sexual abstinence) for at least 30 days after the last dose of the study drug. Negative pregnancy test should be obtained before randomization. The following women are not considered to have childbearing potential: 1) those who have undergone surgical sterilization, including hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy, but excluding bilateral tubal occlusion; 2) age ≥ 50 and post-menopausal as defined by amenorrhea for 12 months or more following cessation of all exogenous hormonal treatments.
  17. Male patients with female partners of childbearing potential who are unwilling to use 2 methods of contraception, one of which must be a barrier method (e.g., condom), for at least 30 days after the last dose of study drug.
  18. Previous exposure to BV100.
  19. Patients who are currently enrolled in or have not yet completed at least 30 days since ending another investigational device or drug trial or are receiving other investigational agents.
  20. Not willing to comply with all study procedures.
  21. Confirmed or suspected severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection based on local standard-of-care assessments available during Screening, unless the suspected A. baumannii pneumonia is diagnosed 14 days or more after the detection of SARS CoV 2.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
To investigate the pharmacokinetic (PK) properties of BV100 co administered with Polymyxin B during 7 to 14 days of treatment in patients with ventilator associated bacterial pneumonia (VABP) | 14 days
  Maximum Observed Plasma Concentration (Cmax) of rifabutin
To investigate the pharmacokinetic properties of BV100 co administered with Polymyxin B during 7 to 14 days of treatment in patients with ventilator associated bacterial pneumonia (VABP) | 14 days
  Area Under the Plasma Concentration-Time Curve (AUC) of rifabutin

SECONDARY OUTCOMES:
To assess the 28 day ACM rates of BV100 plus Polymyxin B compared to best available therapy (BAT) | 28 Days
  28 Day ACM
To assess the 14 day ACM rates of BV100 plus Polymyxin B compared to best available therapy (BAT) | 14
  14 Day ACM
To assess safety and tolerability of BV100 plus Polymyxin B compared to best available therapy (BAT) | 28 days
  Number of Participants with Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Husband, MD, Study Director — BioVersys SAS
Locations (16):
- Georgia (7):
  - Academician Vakhtang Bochorishvili Clinic, Tbilisi
  - Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
  - First University Clinic of Tbilisi State Medical University, Tbilisi
  - Gudushauri National Medical Center, Tbilisi
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center, Tbilisi
  - Number 5 Clinical Hospital, Tbilisi
  - Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic, Tbilisi
- Greece (6):
  - General Hospital of Athens "Evangelismos", Athens
  - University General Hospital "Attikon", Athens
  - General University Hospital of Heraklion, Heraklion
  - General Hospital of Larissa, Larissa
  - University General Hospital of Larissa, Larissa
  - General Hospital of Thessaloniki "Ippokratio", Thessaloniki
- Hungary (3):
  - University of Debrecen Clinical Center, Debrecen
  - University Educational Hospital, Miskolc
  - Fejer County St. Gyorgy University Teaching Hospital, Székesfehérvár